CLINICAL TRIAL: NCT03433534
Title: Study of the Concentration-effect Relationship of Nivolumab in Patients With Kidney or Lung Cancer
Acronym: NIVEAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI17/NIVEAL; 2017-A02788-45 (Other: IdRCB); 2017.12.08 (Other: CPP)
Record Dates: First submitted 2018-01-24; First posted 2018-02-14 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Kidney Cancer; Lung Cancer
Keywords: nivolumab; monoclonal antibody; Opdivo; antineoplastic agent; ELISA; pharmacokinetic
MeSH Terms: conditions — Kidney Neoplasms; Lung Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn to all patients to measure nivolumab concentration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pharmacokinetic of Nivolumab: Patients under nivolumab (Opdivo 10 MG/ML) for the treatment of non small cell lung carcinoma or renal cell carcinoma. Measure of nivolumab residual concentration 14 days after administration of nivolumab and just before the new perfusion.
  Interventions: Other: Pharmacokinetic of Nivolumab

INTERVENTIONS:
Other: Pharmacokinetic of Nivolumab — Nivolumab residual concentration is measured 14 days after administration of nivolumab 3 mg/kg as an intravenous infusion just before the new administration.
  Other Names: Opdivo

SUMMARY:
To assess the relationship between progression free survival of patients treated with nivolumab for metastatic non small cell lung carcinoma or a metastatic renal cell carcinoma and nivolumab blood concentration.

Collection of standard data prospectively.

DETAILED DESCRIPTION:
Nivolumab is a monoclonal antibody used for the treatment of non small cell lung carcinoma and renal cell carcinoma. Huge variability exists between patients treated by nivolumab in terms of efficacy and side effects. Like others monoclonal antibodies, a relation between concentration and effects of nivolumab may exist.

The aim of this study is to assess the relationship between blood concentration of nivolumab and progression free survival, overall survival and side effects on the one hand, and on the other to describe pharmacokinetic of nivolumab

ELIGIBILITY:
Inclusion Criteria:

* Patient with squamous or non squamous non small cell lung cancer stage IV or patient with renal cell carcinoma stage IV
* Patient receiving nivolumab or who will receive nivolumab
* Age ⩾ 18 years old
* OMS stage ≤ 2
* Evaluable disease

Exclusion Criteria:

* Active brain metastasis not treated before by surgery or radiotherapy
* Autoimmune disease
* Patient having objected to the processing of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with nivolumab at CHRU of Tours for squamous or non squamous non small cell lung cancer stage IV or renal cell carcinoma stage IV
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Up to one year
  Association between nivolumab concentration and progression free survival : time from start of nivolumab treatment to progression

SECONDARY OUTCOMES:
Overall survival | Up to one year
  Association between nivolumab concentration and overall survival : time from start of nivolumab treatment to death
Target concentration | 14 days
  Determination of nivolumab concentration associated with clinical benefit (complete response + partial response + stable disease)
Side effects | 14 days
  Association between nivolumab residual concentration and side effects
Nivolumab PK parameters : distribution volume | Baseline up to one year
  Nivolumab residual concentrations will be measured each 14 days until the end of the study (up to one year).
Nivolumab PK parameters : clearance | Baseline up to one year
  Nivolumab residual concentrations will be measured each 14 days until the end of the study (up to one year).

CONTACTS AND LOCATIONS:
Overall Officials: Claude Linassier, Study Director — University Hospital, Tours
Locations (2):
- France (2):
  - Medical oncology department, University Hospital, Tours, Tours
  - Pneumology department, University Hospital, Tours, Tours